CLINICAL TRIAL: NCT03127813
Title: The PAIR Study. Positive Airway Pressure and Intraocular Relationship: IOP Response to a Short-term Application of CPAP
Brief Title: PAIR Study-PAP And IOP Relationship: Study 1
Acronym: PAIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After recruiting just over 50% of target an interim review conclude a larger sample size was highly unlikely to alter the study outcomes
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Hinchingbrooke Hospital NHS Trust (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: P02133
Record Dates: First submitted 2017-04-13; First posted 2017-04-25 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Obstructive Sleep Apnoea; Primary Open Angle Glaucoma
Keywords: glaucoma; OSA; apnoea; intraocular; CPAP; airway; pressure; blindness
MeSH Terms: conditions — Sleep Apnea, Obstructive; Glaucoma, Open-Angle; Glaucoma; Apnea; Blindness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treated glaucoma (Experimental): POAG patients established on treatment
  Interventions: Other: Application of continuous positive airway pressure (CPAP)
- Untreated (Experimental): Newly diagnosed treatment naïve POAG patients
  Interventions: Other: Application of continuous positive airway pressure (CPAP)
- Control (Active Comparator): Control subjects without glaucoma
  Interventions: Other: Application of continuous positive airway pressure (CPAP)

INTERVENTIONS:
Other: Application of continuous positive airway pressure (CPAP) — CPAP will be delivered at 4 different pressure levels (6, 10, 13 and 16cmH2O) in a randomly allocated order

SUMMARY:
Lowering of the pressure in the eye (intraocular pressure, IOP) is the only proven treatment for Primary Open-angle Glaucoma (POAG). However, even effective reduction of IOP by pharmacological or surgical means does not always change the course of the disease or prevent the onset of glaucoma. Some people with POAG also suffer from Obstructive Sleep Apnoea (OSA), an increasingly common sleep disorder which is known to affect heart and blood vessels, and may contribute to glaucoma progression. OSA is treated with Continuous Positive Airway Pressure (CPAP); however using this type of breathing support may raise IOP.

This study aims to establish whether a short-term application of CPAP in awake subjects leads to an increase in IOP. Patients with treated POAG, patients with newly diagnosed untreated POAG and control subjects without glaucoma will be included. CPAP will be applied at several different pressure levels for a total of 2 hours during which IOP and ocular perfusion pressure (OPP) will be measured. If CPAP is shown to raise IOP or alter OPP it could be necessary to assess available alternative treatment options for OSA.

DETAILED DESCRIPTION:
Primary open-angle glaucoma (POAG) is a progressive optic neuropathy characterized by specific optic disc changes and associated visual field defects. Estimated prevalence is 3.0%, making it the leading cause of irreversible blindness worldwide. Intraocular pressure (IOP) is the only proven modifiable risk factor for the development and progression of POAG, but even effective reduction of IOP by pharmacological or surgical means does not always change the course of the disease or prevent some people from developing glaucoma.

OSA is a sleep-related breathing disorder (SBD) caused by complete (apnoea) or partial (hypopnoea) narrowing of the upper airway, resulting in disturbed sleep and intermittent oxygen desaturations. These in turn have negative impact on cardiovascular system and potentially other organs. OSA is treated by continuous positive airway pressure (CPAP) applied by a nasal or a full face mask which maintains patency of the upper airway. CPAP is the first line treatment for moderately severe and severe OSA and, among currently used treatment modalities, it is also the most effective one. The prevalence of OSA continues to increase linked with the rising global incidence of obesity, though many remain undiagnosed. A recent study from the United States estimated that 35% of people between the ages of 50 and 70 years suffer from OSA, and approximately 12% may require treatment.

OSA and OAG are, therefore, two common conditions which may coexist in a significant proportion of patients. In fact, some studies indicate increased prevalence of OAG in patients with OSA, which is in line with a suspected causative role of OSA in glaucoma.

People with OAG and concomitant OSA associated with the relevant symptoms, particularly daytime sleepiness, currently receive standard treatment with CPAP. However, the impact of CPAP on their glaucoma is unknown. There are concerns that CPAP increases IOP, currently the only modifiable factor in glaucoma, though the evidence for this is limited. The exact mechanisms of the possible IOP-raising effect of CPAP are not clear. The favoured hypothesis is CPAP leads to increases in intrathoracic pressure, which in turn raises pressure in the venous circulation and a reduction in the aqueous humour outflow through the episcleral veins and ultimately IOP increase. A similar mechanism is believed to be responsible for IOP elevation in the transition from an upright to supine position in which venous drainage is reduced.

The relationship between the level of pressure used in CPAP treatment and IOP has not been studied. It is unknown if IOP increases in correlated way to CPAP or whether there is no straightforward correlation. If the first is true, application of CPAP only up to a certain pressure level would be safe and perhaps the threshold to use bi-level PAP should be lower in patients with glaucoma. If, however, IOP changes are a matter of individual response to CPAP, perhaps dependent on the severity of OSA or BMI, a routine measurement of the pressure should be performed once CPAP is started. This is currently not a part of standard clinical practice. It is also possible that CPAP set within the usual pressure range does not influence IOP or its effect is not mediated by simple mechanical pressure transmission.

Therefore understanding the influence of CPAP on IOP is important as it may inform the management of people with OSA and concomitant glaucoma. If CPAP is shown to raise IOP or alter ocular perfusion pressure (OPP) to levels that pose clinical risk it will be necessary to assess available alternative treatment options for OSA.

This is a prospective physiological controlled study which will assess IOP response to several different CPAP levels applied for short periods in wakefulness in three groups of people: POAG patients established on treatment (treated glaucoma group), newly diagnosed treatment naïve POAG patients (untreated glaucoma group) and control subjects without glaucoma (control subjects).

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years
* Able to give informed consent and attend for the study visit.

Exclusion Criteria:

* Previous surgical treatment for glaucoma
* Current or recent (within 4 weeks) CPAP or non-invasive ventilation (NIV) use
* History of face mask intolerance
* Any facial lesion preventing safe CPAP mask application
* Allergy to silicone
* Any contraindications to rebound tonometry, including: corneal scarring, microphthalmos, buphthalmos, nystagmus, keratoconus, abnormal central corneal thickness, corneal ectasia, active corneal infection, , and corneal dystrophies.
* Concomitant eye diseases known to affect IOP, including: treated wet age related macular degeneration (ARMD), central retinal vein occlusion (CRVO), branch retinal vein occlusion (BRVO), uveitis and diabetic retinopathy.
* Significant lung disease (including previous pneumothorax, previous or current respiratory failure, severe Chronic Obstructive Pulmonary Disease (COPD), bullous lung disease, difficult to control asthma, acute chest infection)
* Significant heart disease (including heart failure, unstable arrhythmias, pulmonary hypertension)
* Untreated upper gastro-intestinal obstruction
* Acute infectious diseases
* Known or suspected pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | On completion of study visit- 3 hours
  Difference between baseline IOP and IOP on each CPAP level

SECONDARY OUTCOMES:
Relationship between Continuous Positive Airway Pressure (CPAP) level and IOP | On completion of study visit - 3hours
  Correlation between level of CPAP applied and IOP
Minimum CPAP level required to increase IOP | On completion of study visit- 3 hours
  Minimum CPAP level required to increase IOP
Differences in change in IOP between each study group | On completion of study visit - 3 hours
  Differences in IOP change (ΔIOP; IOPCPAP -IOPbaseline) at each CPAP level between the study groups
Relationship between changes in IOP after CPAP with BMI | On completion of study visit - 3 hours
  Correlation between IOP change (ΔIOP; IOPCPAP -IOPbaseline) in response to CPAP with BMI
Relationship between changes in IOP after CPAP with lung volume (Vital Capacity-VC) | On completion of study visit - 3 hours
  Correlation between IOP change (ΔIOP; IOPCPAP -IOPbaseline) in response to CPAP with Vital Capacity
Relationship between changes in IOP after CPAP with glaucoma severity. | On completion of study visit - 3 hours
  Correlation between IOP change (ΔIOP; IOPCPAP -IOPbaseline) in response to CPAP with glaucoma severity

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Wozniak, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Hinchingbrooke Hospital NHS Foundation Trust, Huntingdon, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815
- [Background] Heijl A, Leske MC, Bengtsson B, Hyman L, Bengtsson B, Hussein M; Early Manifest Glaucoma Trial Group. Reduction of intraocular pressure and glaucoma progression: results from the Early Manifest Glaucoma Trial. Arch Ophthalmol. 2002 Oct;120(10):1268-79. doi: 10.1001/archopht.120.10.1268. PMID 12365904
- [Background] Kohler M. Deleterious systemic effects of OSA: how much evidence do we need? Thorax. 2015 Sep;70(9):817-8. doi: 10.1136/thoraxjnl-2015-207247. Epub 2015 Jul 14. No abstract available. PMID 26173952
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Bendel RE, Kaplan J, Heckman M, Fredrickson PA, Lin SC. Prevalence of glaucoma in patients with obstructive sleep apnoea--a cross-sectional case-series. Eye (Lond). 2008 Sep;22(9):1105-9. doi: 10.1038/sj.eye.6702846. Epub 2007 May 4. PMID 17479120
- [Background] Mojon DS, Hess CW, Goldblum D, Fleischhauer J, Koerner F, Bassetti C, Mathis J. High prevalence of glaucoma in patients with sleep apnea syndrome. Ophthalmology. 1999 May;106(5):1009-12. doi: 10.1016/S0161-6420(99)00525-4. PMID 10328405
- [Background] Kiekens S, Veva De Groot, Coeckelbergh T, Tassignon MJ, van de Heyning P, Wilfried De Backer, Verbraecken J. Continuous positive airway pressure therapy is associated with an increase in intraocular pressure in obstructive sleep apnea. Invest Ophthalmol Vis Sci. 2008 Mar;49(3):934-40. doi: 10.1167/iovs.06-1418. PMID 18326715
- [Background] Pepin JL, Chiquet C, Tamisier R, Levy P, Almanjoumi A, Romanet JP. Frequent loss of nyctohemeral rhythm of intraocular pressure restored by nCPAP treatment in patients with severe apnea. Arch Ophthalmol. 2010 Oct;128(10):1257-63. doi: 10.1001/archophthalmol.2010.220. PMID 20937994
- [Background] Becker H, Grote L, Ploch T, Schneider H, Stammnitz A, Peter JH, Podszus T. Intrathoracic pressure changes and cardiovascular effects induced by nCPAP and nBiPAP in sleep apnoea patients. J Sleep Res. 1995 Jun;4(S1):125-129. doi: 10.1111/j.1365-2869.1995.tb00201.x. PMID 10607188